CLINICAL TRIAL: NCT02525198
Title: A Randomised Controlled Trial in 'At Risk' Humans Investigating the Cognitive Benefits of a Combined Flavonoid/Fatty Acid Intervention and Underlying Mechanisms of Action: The COGNITIVE AGING NUTRITION and NEUROGENESIS (CANN) Trial
Brief Title: The Cognitive Ageing Nutrition and Neurogenesis (CANN) Trial
Acronym: CANN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Swinburne University of Technology (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21647
Record Dates: First submitted 2015-05-11; First posted 2015-08-17 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment; Subjective Memory Impairment
Keywords: Mild cognitive impairment; Subjective memory impairment; Dementia; Flavonoids; Fatty acids; Cognition; Gut microflora
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo group: 12 month daily ingestion of placebo oil and flavonoid-poor matched extract
  Interventions: Dietary Supplement: Placebo
- fatty acid/flavonoid blend (Experimental): Experimental group: 12 month daily ingestion of 1.5 g EPA+DHA and 500 mg flavonoids
  Interventions: Dietary Supplement: fatty acid/flavonoid blend

INTERVENTIONS:
Dietary Supplement: fatty acid/flavonoid blend — see arm description
  Arms: fatty acid/flavonoid blend
Dietary Supplement: Placebo — see arm description
  Arms: Placebo

SUMMARY:
There is a dearth of research which takes a multi-compound approach to dietary interventions, in humans, aimed at improving outcome measures of cognition. Animal research in particular points towards fatty acids and flavonoids having a potentiating effect on each other, and possibly even being synergistic. Thus, study products will be administered in the present trial comprising both of these compounds, with a view to investigating their potential effects on cognition in older adults with mild cognitive impairment (MCI) or subjective memory impairment (SMI).

DETAILED DESCRIPTION:
240 participants, aged 55 or above, will be recruited (120 Norwich, 120 Melbourne; to include both MCI and SCI participants).

Participants will be asked to take the study food each day for 12 months, and to come to the clinical assessment unit on 3 occasions, at baseline, 3 months and 12 months, to complete a cognitive task battery such that their performance may be investigated in the context of the intervention.

Urine, blood and faecal samples will be collected and magnetic resonance imaging (MRI) will be applicable to half of each population (i.e to 60 MCI and 60 SCI, 30 of each at Norwich and Melbourne).

ELIGIBILITY:
Inclusion Criteria:

* Male and female, aged ≥ 55 years
* Mild cognitive impairment (MCI) or subjective memory impairment (SMI) with no indication of clinical dementia or depression
* Willing and able to provide written informed consent.
* Understands and is willing and able to comply with all study procedures.
* Fluent in written and spoken English.
* In good general health including blood biochemical, haematological and urinalysis within the normal range at screening (as judged by the clinical advisor)
* Normal, or corrected to normal vision and hearing
* Right handed, for MRI
* Stable use of any prescribed medication for at least four weeks

Exclusion Criteria:

* Diagnosis of Alzheimer's disease (AD) or other form of dementia or significant neurological disorder
* Parent or sibling who developed premature dementia <60y (suggestive of a familial monogenic form of cognitive decline)
* Past history or MRI evidence of brain damage including significant trauma, stroke, learning difficulties or serious neurological disorder, including loss of consciousness > 24 hours
* History of alcohol or drug dependency within the last 2 years
* Other clinically diagnosed psychiatric disorder likely to affect the cognitive measures (as judged by clinical adviser)
* Existing diagnosed gastrointestinal disorders likely to impact on absorption of flavonoids and fatty acids (as judged by clinical adviser)
* Major cardiovascular event, e.g. myocardial infarction or stroke, in the last 12 months
* Carotid stents or severe stenosis
* Known allergy to fish or any other component in the intervention supplements
* Existing medical conditions likely to affect the study measures (as judged by clinical adviser)
* Uncontrolled hypertension (Systolic Blood Pressure (SBP) >140mmHg, Diastolic Blood Pressure (DBP) >90mmHg)
* BMI >40kg/m2

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Number of false positive responses during the picture recognition task of the CDR Computerized Cognitive Assessment System | 12 months
  The CDR Computerized Cognitive Assessment System will be used to measure the cognitive effects of the treatments. The battery is sensitive to bidirectional cognitive change including trials in MCI, dementia and SMI. There is strong converging evidence that one particular aspect of performance, namely the number of false positive responses during a picture recognition task, is particularly sensitive to hippocampal integrity (based on activation of the dentate gyrus during the task, and specific decrements in conditions associated with poorer hippocampal function). This will form the primary outcome in this study.

SECONDARY OUTCOMES:
Hippocampal volume | 12 months
  To be measured on magnetic resonance imaging
Gut microflora speciation and metabolism | 12 months
  Measured in faecal samples. By extension, we also seek to consider the contribution of the microflora to cognition function and its response to treatment.
Association between baseline APOE status and number of false positive responses during the picture recognition task of the CDR Computerized Cognitive Assessment System | 12 months
  We will assess the impact of intervention in respect to presence or absence of APOE 4 gene across participants, which is a risk factor for dementia.
Circulating biomarkers of cognition | 12 months
  Biomarkers to include BDNF, β-amyloid, plasma lipids, inflammatory markers, nitric oxide and fatty acids, flavonoids and their metabolites (plasma and urine)
Circulating biomarkers of cardiovascular health | 12 months
  Biomarkers to include BDNF, β-amyloid, plasma lipids, inflammatory markers, nitric oxide and fatty acids, flavonoids and their metabolites (plasma and urine)
Language ability on the Boston Naming Test | 12 months
  Allows for categorization according to cognitive status (mild cognitive impairment, dementia, subjective memory impairment)
Visuospatial ability on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Figure Copy test | 12 months
  Allows for categorization according to cognitive status (mild cognitive impairment, dementia, subjective memory impairment)
Attention ability on the Digit Span task | 12 months
  Allows for categorization according to cognitive status (mild cognitive impairment, dementia, subjective memory impairment)
Executive function on the Trail Making Task | 12 months
  Allows for categorization according to cognitive status (mild cognitive impairment, dementia, subjective memory impairment)
Cerebrovascular blood flow | 12 months
  To be measured on spectroscopy
Measurement of blood brain barrier permeability | 8 minutes
  Allows testing of the hypothesis that the test food will help improve BBB permeability through its action on endothelial function. Six axial slices will be measured every 1.34 seconds for 8 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Minihane, PhD, Principal Investigator — Department of Nutrition, University of East Anglia, Norwich, U.K.; Andrew Scholey, PhD, Principal Investigator — Centre for Human Psychopharmacology, Swinburne University of Technology; Neal J Cohen, PhD, Principal Investigator — Beckman Institute, University of Illinois
Locations (3):
- Beckman Institute, University of Illinois, Urbana, Illinois, United States
- Centre for Human Psychopharmacology, Swinburne Univerity of Technology, Melbourne, Victoria, Australia
- Department of Nutrition, University of East Anglia, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Vauzour D, Scholey A, White DJ, Cohen NJ, Cassidy A, Gillings R, Irvine MA, Kay CD, Kim M, King R, Legido-Quigley C, Potter JF, Schwarb H, Minihane AM. A combined DHA-rich fish oil and cocoa flavanols intervention does not improve cognition or brain structure in older adults with memory complaints: results from the CANN randomized, controlled parallel-design study. Am J Clin Nutr. 2023 Aug;118(2):369-381. doi: 10.1016/j.ajcnut.2023.06.008. Epub 2023 Jun 12. PMID 37315924
- [Derived] Irvine MA, Scholey A, King R, Gillings R, Vauzour D, Demichele SJ, Das T, Wesnes KA, Sutton BP, Cassidy A, Pipingas A, Potter JF, Johnson G, White D, Larsen R, Cohen NJ, Minihane AM. The Cognitive Ageing, Nutrition and Neurogenesis (CANN) trial: Design and progress. Alzheimers Dement (N Y). 2018 Sep 5;4:591-601. doi: 10.1016/j.trci.2018.08.001. eCollection 2018. PMID 30426067